CLINICAL TRIAL: NCT03796897
Title: Supplementation of a Leucine-Enriched Dairy Protein Blend: Chronic and Acute Metabolic Responses in Young Men and Women
Brief Title: Supplementation of a Leucine-enriched Protein Blend
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Stuart Phillips, Professor, McMaster University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 5706
Record Dates: First submitted 2019-01-07; First posted 2019-01-08 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Dietary Modification; Diet Habit
MeSH Terms: conditions — Feeding Behavior | interventions — P3H1 protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Leucine-enriched protein + exercise (Experimental): whey protein- hydrolyzed whey protein-micellar casein blend (50:43:7 whey:hydrolyzed-whey:casein), vitamin D, and free leucine
  Interventions: Dietary Supplement: Leucine-enriched protein
- Habitual diet + exercise (Sham Comparator): habitual diet only
  Interventions: Behavioral: Habitual diet only

INTERVENTIONS:
Dietary Supplement: Leucine-enriched protein — Supplement contains 16g of protein given twice per exercise session (4 total exercise sessions)
  Arms: Leucine-enriched protein + exercise
Behavioral: Habitual diet only — Habitual diet only (no supplementation) for 4 exercise sessions
  Arms: Habitual diet + exercise

SUMMARY:
It is well known that dietary protein transiently stimulates muscle protein synthesis (MPS) whereby changes in MPS in response to feeding may be regulated by specific downstream target proteins of mammalian target of rapamycin signaling, such as S6K1, rpS6, and eIF2B. A meal deficient in protein, however, does not increase the rate of MPS because a rise in the bioavailability of amino acids does not occur. In addition, the source of dietary proteins has been shown to impact postprandial blood levels of amino acids. The concept that certain types of proteins are "fast acting" or "slow acting" has been shown to affect the postprandial profile of amino acids appearing in the systemic circulation. Native whey and micellar casein are both dairy proteins that contain a similar amount of essential (EAA), but blood EAA levels increase faster and to a higher level after the consumption of whey protein. Differences in gastric emptying, digestion and absorption kinetics between micellar casein and native whey are the underlying factors. Nonetheless, micellar casein protein has been shown to protract MPS in humans. Despite the significant amount of information gained with respect to both of these protein sources, the effects of combinatorial formulations on the postprandial profile of amino acids appearing in the blood is less well known.

DETAILED DESCRIPTION:
In a cross-over, randomized controlled trial, 10 healthy young participants (5 men and 5 women) will be recruited to undergo exercise resistance training randomized to habitual diet or habitual diet and supplementation (2 x per training session). For two of the training sessions the investigators will utilize a uni-lateral resistance exercise model to identify the acute effects of exercise and exercise + supplementation on the integrated rate of myofibrillar MPS within subject. This model enhances statistical power and eliminates between-subject differences impacting our outcomes. Throughout the study participants will record their macronutrient dietary intake. In addition, baseline body composition will be assessed with dual-energy x-ray absorptiometry.

Visit 1 (Day -7): Familiarization, strength testing and baseline body composition One week before the exercise trial, the investigators will ask participants to visit McMaster University to undergo a familiarization session with the exercise equipment and to perform 3-5 repetition maximum strength testing. This will allow the investigators to calculate the resistance (weight) participants will lift in their upcoming training sessions. The investigators will also perform a body composition scan using a dual-energy x-ray absorptiometry (DXA), assess participants' height and weight, and administer daily food logs with instructions to assess their habitual diet.

Visit 2 (Day 0): D2O administration and resting blood and saliva sampling One week after the familiarization visit, the investigators will ask participants to come to McMaster University in a fasted state and receive a dose of doubly labelled water D2O equal to 0.8mLs/kgBW and every hour for 3 hours after providing a blood and saliva sample. D2O is a safe, and widely used stable isotope, used to effectively measure the rate at which participants' muscle grow.

Visits 3 and 7 (Days 1 and 7): Resistance training program and muscle biopsy On these days participants will come to the lab in the morning following their habitual diet routine and will have a resting biopsy, blood and saliva samples taken. Next, participants may be asked to consume the supplement but will be asked to drink a small amount of D2O. Finally, participants will perform a combination resistance style exercise training session and immediately following training may be asked to consume the supplement.

Visit 4, 5, 8 & 9 (Days 2, 3, 8, 9): Resistance training program On these days participants will come to the lab in the morning following their habitual diet routine and have a saliva sample taken. Next, participants may be asked to consume the supplement but will be asked to drink a small amount of D2O. Finally, participants will perform a combination resistance style exercise training session and immediately following training participants may be asked to consume the supplement.

Visits 6 and 10 (Days 4 and 10): Uni-lateral acute training session and muscle biopsy On these days participants will come to the lab in the morning following their habitual diet routine. First, participants may be asked to consume the supplement immediately before performing a uni-lateral acute resistance training session. Participants will be asked to drink a small amount of D2O but only during Visit 6 (Day 4). Immediately following training, participants may be asked to consume the supplement. One hour following exercise participants will have a muscle biopsy, blood and saliva samples taken.

Days 5 and 6 (see attached study timeline): Washout period The investigators will ask that participants drink one aliquot of D2O on day 5 and one aliquot of D2O on day 6. One hour after participants drink the aliquot of D2O the investigators ask that participants take their own saliva sample at home (D2O aliquots and a sampling kit will be provided with instructions).

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 18-29 years (inclusive)
* Be able to maintain a habitual diet, physical activity patterns, and body mass throughout the trial
* Be in general good health
* Be able to participate in resistance training and aerobic training
* Understand the study procedures and sign this form providing informed consent to participate in the study
* Be able to consume a protein bar in the allotted time frame of 10 minutes

Exclusion Criteria:

* Smoker
* Excessive alcohol consumption (more than 21 units of alcohol / week; 1 unit of alcohol is approximately 25 mL of spirits (40% alcohol), 250 mL of beer (4% alcohol) or 75 mL of wine (13% alcohol))
* Have health problems such as: renal or gastrointestinal disorders, metabolic disease, heart disease, vascular disease, rheumatoid arthritis, diabetes, poor lung function, uncontrolled blood pressure, dizziness, thyroid problems, or any other health conditions for which you are being treated that might put you at risk for this study
* Have a known or suspected allergy to local anesthetics such as lidocaine
* Have a dairy protein allergy
* Participation in another nutrition or exercise research study
* Do not understand English or have a condition the PI believes would interfere with a participants' ability to provide informed consent, comply with the study protocol, or which might confound the interpretation of the study results or put someone at undue risk
* Use of medications known to affect protein metabolism (i.e. corticosteroids, or prescription strength acne medications)
* Consuming a vegan diet
* Use of an investigational drug product or nutraceutical within the last 30 days
* Any concurrent medical, orthopedic, or psychiatric condition that, in the opinion of the Investigators, would compromise the ability to comply with the study requirements

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Integrated Muscle Protein Synthetic Rate | 10 days
  oral deuterium consumption: Isotope protocol (See ref., PMID 23821570)

CONTACTS AND LOCATIONS:
Locations (1):
- Exercise Metabolism Research Laboratory, McMaster Univeristy, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Koopman R, Crombach N, Gijsen AP, Walrand S, Fauquant J, Kies AK, Lemosquet S, Saris WH, Boirie Y, van Loon LJ. Ingestion of a protein hydrolysate is accompanied by an accelerated in vivo digestion and absorption rate when compared with its intact protein. Am J Clin Nutr. 2009 Jul;90(1):106-15. doi: 10.3945/ajcn.2009.27474. Epub 2009 May 27. PMID 19474134
- [Result] Koopman R, Walrand S, Beelen M, Gijsen AP, Kies AK, Boirie Y, Saris WH, van Loon LJ. Dietary protein digestion and absorption rates and the subsequent postprandial muscle protein synthetic response do not differ between young and elderly men. J Nutr. 2009 Sep;139(9):1707-13. doi: 10.3945/jn.109.109173. Epub 2009 Jul 22. PMID 19625697
- [Result] Moore DR, Robinson MJ, Fry JL, Tang JE, Glover EI, Wilkinson SB, Prior T, Tarnopolsky MA, Phillips SM. Ingested protein dose response of muscle and albumin protein synthesis after resistance exercise in young men. Am J Clin Nutr. 2009 Jan;89(1):161-8. doi: 10.3945/ajcn.2008.26401. Epub 2008 Dec 3. PMID 19056590
- [Result] Katsanos CS, Kobayashi H, Sheffield-Moore M, Aarsland A, Wolfe RR. A high proportion of leucine is required for optimal stimulation of the rate of muscle protein synthesis by essential amino acids in the elderly. Am J Physiol Endocrinol Metab. 2006 Aug;291(2):E381-7. doi: 10.1152/ajpendo.00488.2005. Epub 2006 Feb 28. PMID 16507602
- [Result] Luiking YC, Abrahamse E, Ludwig T, Boirie Y, Verlaan S. Protein type and caloric density of protein supplements modulate postprandial amino acid profile through changes in gastrointestinal behaviour: A randomized trial. Clin Nutr. 2016 Feb;35(1):48-58. doi: 10.1016/j.clnu.2015.02.013. Epub 2015 Mar 5. PMID 25790724
- [Result] Tipton KD, Elliott TA, Cree MG, Wolf SE, Sanford AP, Wolfe RR. Ingestion of casein and whey proteins result in muscle anabolism after resistance exercise. Med Sci Sports Exerc. 2004 Dec;36(12):2073-81. doi: 10.1249/01.mss.0000147582.99810.c5. PMID 15570142
- [Result] Boirie Y, Dangin M, Gachon P, Vasson MP, Maubois JL, Beaufrere B. Slow and fast dietary proteins differently modulate postprandial protein accretion. Proc Natl Acad Sci U S A. 1997 Dec 23;94(26):14930-5. doi: 10.1073/pnas.94.26.14930. PMID 9405716
- [Result] MacDonald AJ, Small AC, Greig CA, Husi H, Ross JA, Stephens NA, Fearon KC, Preston T. A novel oral tracer procedure for measurement of habitual myofibrillar protein synthesis. Rapid Commun Mass Spectrom. 2013 Aug 15;27(15):1769-77. doi: 10.1002/rcm.6622. PMID 23821570
- [Derived] Lim C, Traylor DA, McGlory C, Joanisse S, McKendry J, Grewal T, Mcleod JC, Prior T, Nunes EA, Lees M, Phillips SM. Increased protein intake derived from leucine-enriched protein enhances the integrated myofibrillar protein synthetic response to short-term resistance training in untrained men and women: a 4-day randomized controlled trial. Appl Physiol Nutr Metab. 2022 Nov 1;47(11):1104-1114. doi: 10.1139/apnm-2022-0164. Epub 2022 Sep 20. PMID 36126327